CLINICAL TRIAL: NCT02194660
Title: Fragility Fracture Liaison Service Project
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201311048RINC
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Osteoporosis; Fracture
Keywords: Fractures Liaison Service; Osteoporosis; Fracture; Medication adherence
MeSH Terms: conditions — Osteoporosis; Fractures, Bone; Medication Adherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- M- main hospital: Patient enrolled in the main hospital
- B- Beihu branch: Patients enrolled in the Beihu branch

SUMMARY:
Aims: to Establish the FLS services at the National Taiwan University Hospital (NTUH) and its Beihu Branch (BB).

Method: From Jan., 2014, two related fracture liaison services (FLSs) following the 13 'Capture the Fracture Best Practice Standards' were implemented at the National Taiwan University Hospital (NTUH) health care system. The main hospital (MH) program enrolled patient with 1) new hip fracture 2) newly identified radiographic vertebral fractures or 3) clinical vertebral fractures from both inpatients and outpatients. The Beihu branch (BB) program enrolled only the later two types of patients from outpatients. During the whole study period, two programs planed to enroll 600 fracture patients. Each patient would be assessed at baseline, and every 4 month for at least one year.

DETAILED DESCRIPTION:
Background:The Asia Fracture Gap Taiwan Study (AFGTS) showed that among fragility fracture sufferers, only 1/4 of them underwent bone mineral density (BMD) tests and 1/3 of them received treatments for osteoporosis. Secondary fragility fracture prevention services are needed to improve the care gaps

. Aims: to Establish the FLS services at the National Taiwan University Hospital (NTUH) and its Beihu Branch (BB).

Method: The FLS was designed following the 13 'Capture the Fracture Best Practice Standards'. The National Taiwan University Hospital (NTUH) institutional review board approved the study in Jan., 2014. Patients were eligible to be enrolled into the main hospital (MH) service if they had

1. new hip fracture in orthopedic ward
2. newly identified radiographic vertebral fractures from plan films in geriatric ward or
3. clinical vertebral fractures in outpatient clinics.

Patients in outpatient clinics of BB were eligible to be enrolled if they had (1) clinical vertebral fractures or (2) newly identified asymtomatic radiological vertebral fractures by a routine weekly review of every plan film of thoracic or lumbar spine regardless of the reason for it.They were excluded from the service if they had life expectancy shorter than 2 years of life or not be able to complete study assessments for communication or cognitive problems.

Osteoporosis-related assessments, treatments, consultations on diet, medications, exercise, fall prevention were given mainly by care managers. A system is set up to remind patients to take their medications at home or to return to clinic for regular injections of medications. Follow up assessments included adherence to education instructions, medications, fall and fracture incidences. During the whole study period, we planed to enroll 600 fracture patients. Each patient would be assessed at baseline, and every 4 months last for two years.

Anticipated results:

Establish domestic FLS model and database Publish preliminary results at the 2014 the IOF 5th Regionals Asia Pacific Meeting in Taipei in November.

Participating physicians and care managers will learn new skills in managing osteoporosis patients.

Application for Best Practice Recognition for the IOF Capture the Fracture Campaign

Preliminary results:

We have enrolled 371 eligible patients into FLS services. From the NTUH program, BMD tests were completed within 8 weeks for over 90% of participants. Also, anti-osteoporosis medication (AOMs) were prescribed to about 90% of participants eligible for National Health Insurance reimbursements.

In 2014, National Taiwan University Hospital (NTUH) and its BeiHu Branch (BB) were awarded the gold medal and silver medal accredited best practice programs from the 'Capture the Fracture' campaign from International Osteoporosis Foundation, respectively.

Our preliminary results were presented at annual scientific meeting of the Taiwanese Osteoporosis Association, at Madrid, Spain, and the IOF 5th Regionals Asia Pacific Meeting in Taipei, Taiwan, and the World Congress on Osteoporosis, Osteoarthritis and Musculoskeletal Diseases, at Milan, Italy.

ELIGIBILITY:
Inclusion Criteria: (Main hospital)

* age >=50 years and
* new hip fracture in orthopedic ward
* newly identified radiographic vertebral fractures from plan films in geriatric ward
* clinical vertebral fractures in outpatient clinics Inclusion criteria (Beihu branch, only outpatients)
* age >=50 years and
* newly identified radiographic vertebral fractures from plan films
* clinical vertebral fractures

Exclusion Criteria:

* fracture is sufer from trauma or cancer
* atypical fractures
* Life expectancy less than 2 years or can't be assessed for communication or cognitive problems
* patient in other medication clinical trials

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: new fragility fracture
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-12-28 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density test within 8 weeks of enrollments | 8 weeks
  Capture the fracture campaign provide 13 best practice standards. The above mentioned index is the limiting factor for many osteoporosis related managements after fracture. We decided to use this as the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital Chu-Tung Branch
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No